CLINICAL TRIAL: NCT00865982
Title: Multicenter, Open Lable Phase II Study to Evaluate the Safety and Efficacy of a Perioperative Chemotherapy With Docetaxel, Cisplatin and Capecitabine in Patients With Gastric Adenocarcinoma, Adenocarcinoma of the Gastro-esophageal Junction or the Distal Esophagus
Brief Title: Study to Evaluate Safety and Efficacy of Perioperative Chemotherapy With Docetaxel, Cisplatin and Capecitabine (DCX) in Patients With Gastro-esophageal Cancer
Acronym: DCXAIOCHARITE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Roche Pharma AG (Industry); Sanofi (Industry)
Responsible Party: Dr. med. Peter Thuss-Patience, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudract-CT-2008-001849-26
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Gastric Cancer; Esophageal Cancer
Keywords: adenocarcinoma of the stomach, gastro-esophageal junction or distal esophagus; gastric cancer; esophageal cancer; gastro-esophageal junction; docetaxel; capecitabine; cisplatin; perioperative chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Docetaxel; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, Capecitabine — 3 preoperative cycles with Docetaxel 75 mg/m² d1 Cisplatin 60 mg/m² d1 Capecitabine 1875 mg/m²/day d1-14 repeated every 3 weeks
  followed by resection
  and 3 postoperative cycles with Docetaxel 75 mg/m² d1 Cisplatin 60 mg/m² d1 Capecitabine 1875 mg/m²/day d1-14 repeated every 3 weeks.

SUMMARY:
In this study, patients with adenocarcinoma of the stomach, gastro-esophageal junction or the distal esophagus who seem operable with curative intent according to oncological and surgical assessment are treated with 3 preoperative cycles of DCX (Docetaxel, Cisplatin, Capecitabine) followed by surgical resection, followed by 3 postoperative cycles of DCX.

DETAILED DESCRIPTION:
Perioperative chemotherapy has been shown to significantly improve the R0 resection rate, the disease free survival and the overall survival in patients with adenocarcinoma of the distal esophagus, the gastro-esophageal junction and the stomach. Therefore perioperative chemotherapy is the new therapeutic standard (Cunningham NEJM 2006, MRC, Lancet 2002, Boige ASCO 2007). The best evaluated regime is the combination of Epirubicin, Cisplatin and 5-FU (ECF) (Cunningham, NEJM 2007). Cisplatin and 5-FU seem to be the most important components forming the backbone of this regime (Boige ASCO 2007).

Docetaxel is a new and highly active agent in gastric cancer. In a randomized phase II study the dual combination of Docetaxel and 5-FU seemed to show similar activity as ECF, administered as first line palliative treatment (Thuss-Patience, JCO, 2005). The three drug combination Docetaxel, Cisplatin, 5-FU has significantly superior efficacy than a combination of Cisplatin und 5-FU, superior quality of life and significantly superior overall survival (Van Cutsem, JCO 2007).

It has been shown that Capecitabine the oral prodrug of 5-FU is similarly active as 5-FU and can replace intravenous 5-FU in combination with Cisplatin in the treatment of gastric cancer. Capecitabine therefore is FDA approved for gastric cancer (Cunningham, ASCO 2006, Kang ASCO 2006).

It seems reasonable to optimize perioperative chemotherapy by including modern chemotherapeutics. The old standard ECF may be improved by integrating Docetaxel und Capecitabine. By adding Docetaxel to the Cisplatin / flouropyrimidin backbone the efficacy of the regime may be improved. The replacement of 5-FU by Capecitabine may improve patients´ convenience and possibly effectiveness of the combination. Therefore the 3 drug combination of Docetaxel, Cisplatin, Capecitabin (DCX) seems to be a highly promising regime regarding effectiveness and convenience.

In this study patients with adenocarcinoma of the stomach, gastro-esophageal junction or the distal esophagus who seem operable with curative intent according to oncological and surgical assessment are treated with 3 preoperative cycles of DCX followed by surgical resection, followed by 3 postoperative cycles of DCX.

The first application of study medication has to be within 21 days of tumour assessment. There will be 3 preoperative cycles every 3 weeks. The experimental perioperative regime evaluated in this study will be Docetaxel/Cisplatin/Capecitabine DCX (75/ 60/ 1875 mg/m2).The operation will be performed 3 to 6 weeks after the end of the third preoperative chemotherapy cycle (counted from day 21 of cycle 3).

Postoperative chemotherapy will start within 6 - 12 weeks after the operation. 3 weeks after the end of the last chemotherapy the final investigation (end of study visit) will be done.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated consent
* Age between minimum 18 and maximum 75 years
* Primary diagnosis of histologically proven adenocarcinoma of the stomach, the gastro-esophageal junction or an adenocarcinoma of the lower third of the esophagus
* Stage II-III, which is in TNM-staging: T3-4, N0-3, M0 or T2, N1-3, M0 or T1, N2, M0. (equivalent to clinical staging uT3-4NXM0, uT1-2N+M0)
* Intended curative resection according to evaluation of an experienced surgeon
* Karnofsky-performance-index > 70%
* Negative pregnancy blood test at screening but not earlier than 72 hours prior to start of chemotherapy for women with child bearing potential
* Adequate haematologic function and liver and renal function: neutrophils > 1,5 x 109/L; thrombocytes > 100 x 109/L; haemoglobin > 10 g/dl, creatinine clearance > 60 ml/min (calculated according to Cockroft and Gault), total bilirubin < 1,0 x UNL; AST and ALT < 1,5 x UNL, AP < 2,5 x UNL
* Complete staging within 3 weeks prior to start of treatment (CT-scan of thorax and abdomen, endosonography, gastroscopy)
* Ability to keep appointments and follow the study protocol
* By CT-scan, endoscopy or endosonography measurable or evaluable disease

Exclusion Criteria:

* Former therapy of gastro-esophageal cancer (operation, chemo- or radiotherapy)
* Diagnosis of another cancer in the last 5 years prior to study entry which has not been cured by operation only (exception in-situ-carcinoma of the cervix or cured non-melanomatose skin cancer)
* Known dihydropyrimidine-dehydrogenase (DPD)-deficiency
* Known contraindication to the planned chemotherapeutics
* Presence of distant metastases
* Anamnestic known serious disease or other concomitant diseases that affect participation in this study, such as:

  * Instable cardiac disease: symptomatic heart failure, symptomatic coronary artery disease, ventricular cardiac arrhythmia not well controlled with medication, myocardial infarction or resuscitation within 6 month before study
  * Active infection necessitating systemic therapy or uncontrolled infection
  * Interstitial lung diseases (for example: pneumonitis or fibrosis of the lung) and indication for interstitial lung disease in chest x-ray or CT-scan respectively
  * Active inflammatory bowel disease or other bowel diseases which provoke chronic diarrhea (defined as > 4 bowel movements per day)
  * Neurological or psychiatric disease including dementia, epilepsy or untreated, symptomatic brain metastases
  * Limited hearing ability
* Presence of upper GI obstruction, leading to inability to swallow ground tablets
* Presence of acute or chronic systemic infection
* Presence of a bowel obstruction within the last 30 days
* Pregnant or lactating women or women with child bearing potential and men without adequate contraception (high effective contraception, defined as Pearl Index < 1) like birth control pill, hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), realized sterilization or sexual abstinence during the study and at least for 3 months after the last infusion
* Any other situation which may lead to an unacceptable high risk for the patient, when he participates in the study
* Parallel treatment in another clinical study or prior participation in this study
* Treatment with any other therapy against the tumor or any parallel radiation
* Parallel treatment with Sorivudine or an chemically related substance like for example Brivudin
* Symptomatic peripheral neuropathy NCI-CTCAE degree > 2
* Intolerance to the study medication or their galencic ingredients or against 5-FU
* Detention in a psychiatric unit or imprisonment (AMG §40 Abs. 1 Nr. 4)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
R0-resection rate | After 3 cycles of preoperative chemotherapy (3 month)

SECONDARY OUTCOMES:
Remission rate according to diagnostic imaging techniques | After 3 cycles of preoperative chemotherapy (3 month)
Pathological remission rate | After 3 cycles of preoperative chemotherapy (3 month)
Operative and postoperative complication rate | Within 30 days after surgery
Resectability rate | After 3 cycles of preoperative chemotherapy (3 month)
Rate of local recurrences and metastasis
Toxicity
30-day mortality | After date of surgery
Overall survival
Overall survival rate | 1,2,3 and 5 years
Event free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thuss-Patience, Dr. med., Study Chair — Charite University, Berlin, Germany
Locations (9):
- Germany (9):
  - HELIOS-Klinik Bad Saarow, Bad Saarow
  - Klinik für Hämatologie, Onkologie und Tumorimmunologie, Charite Campus Buch, Berlin
  - Medizinische Klinik mit Schwerpunkt Gastroenterologie, Infektiologie und Rheumatologie, Charite Campus Benjamin-Franklin, Berlin
  - Medizinische Klinik mit Schwerpunkt Hämatologie und Onkologie, Charite Campus Virchow Klinikum, Berlin
  - Klinik für Innere Medizin Abteilung Hämatologie/Onkologie, Städtisches Klinikum Dessau, Dessau
  - Universitätsklinik und Poliklinik für Innere Medizin IV, Martin Luther Universität Halle-Wittenberg, Halle
  - II. Medizinische Klinik und Poliklinik, Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Internistische Onkologie/ Hämatologie, Städtisches Krankenhaus St. Georg, Leipzig
  - 3. Medizinische Klinik, Onkologisches Zentrum, Universitätsklinikum Mannheim, Mannheim

REFERENCES:
- [Derived] Thuss-Patience PC, Hofheinz RD, Arnold D, Florschutz A, Daum S, Kretzschmar A, Mantovani-Loffler L, Bichev D, Breithaupt K, Kneba M, Schumacher G, Glanemann M, Schlattmann P, Reichardt P, Gahn B. Perioperative chemotherapy with docetaxel, cisplatin and capecitabine (DCX) in gastro-oesophageal adenocarcinoma: a phase II study of the Arbeitsgemeinschaft Internistische Onkologie (AIO)dagger. Ann Oncol. 2012 Nov;23(11):2827-2834. doi: 10.1093/annonc/mds129. Epub 2012 Jun 24. PMID 22734012